CLINICAL TRIAL: NCT06394349
Title: Platelet-rich Plasma Intradermal Injection in Addition to 308 nm Excimer Light in the Treatment of Stable Acral Vitiligo: A Prospective Randomized Placebo-controlled Study
Brief Title: Platelet-rich Plasma Intradermal Injection Combined With 308 nm Excimer Light for Treating Stable Acral Vitiligo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yijian Zhu (Other)
Responsible Party: Sponsor-Investigator, Yijian Zhu, Resident Physician, Huashan Hospital
Organization: Huashan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023M-013
Record Dates: First submitted 2024-04-24; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Vitiligo
Keywords: Acral vitiligo; Platelet-rich plasma; 308 nm excimer light
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP+308nm (Experimental): The observation group received PRP intradermal injections (0.5cm apart, 0.02ml injected) once a month and 308 nm excimer phototherapy twice a week for 6 consecutive months.
  Interventions: Combination Product: PRP+308nm
- NS+308nm (Placebo Comparator): The control group received the same frequency of saline injections (0.5cm apart, 0.02ml injected) and phototherapy for 6 consecutive months.
  Interventions: Combination Product: NS+308nm

INTERVENTIONS:
Combination Product: PRP+308nm — PRP+308nm
  Arms: PRP+308nm
Combination Product: NS+308nm — NS+308nm
  Arms: NS+308nm

SUMMARY:
The goal of this clinical trial is to learn if platelet-rich plasma (PRP) works to treat acral stable vitiligo in adults. It will also learn about the safety of platelet-rich plasma. The main questions it aims to answer are:

* Does PRP combined with 308 nm excimer phototherapy improve the efficacy compared to 308 nm excimer light alone in the treatment of vitiligo of the extremities?
* What medical problems do participants have when taking PRP intradermal injections?

Researchers will compare PRP to a placebo (a look-alike substance that contains no drug) to see if PRP works to treat acral vitiligo.

Participants will:

* Receive PRP intradermal injections once a month and 308 nm excimer phototherapy twice a week, or the same frequency of saline injections and phototherapy for 6 consecutive months
* Visit the clinic once every 1 month for evaluations
* Keep a diary of their symptoms or side effects during follow-up

DETAILED DESCRIPTION:
Vitiligo is an acquired skin disorder characterized by depigmented macules, and one of the conventional treatment principles is to promote the differentiation of stem cells at the follicular bulge into melanocytes, but vitiligo of the extremities is clinically difficult to repigmentation and resistant to treatment due to its lack of hair follicles. Platelet-rich plasma (PRP) is a concentrated platelet plasma obtained by in vitro isolation of autologous whole blood, and its effect on repigmentation of vitiligo at the extremities and the potential mechanism remain unclear. The investigators investigated the efficacy of PRP on acral vitiligo by a single-center, prospective, self-controlled clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-segmental vitiligo stable for more than half a year;
* At least 1 separate stable lesion on each of the dorsum of the right and left hands, proximal fingers, distal fingers and palms;
* The area of white spots is less than 10 % of the total body surface area and more than 1 % of the total body surface area;
* Those who have not received systemic treatment of vitiligo and phototherapy or related treatments within 1 month ≥ 1 year without significant efficacy;
* Voluntary signing of informed consent.

Exclusion Criteria:

* Pregnant and lactating women;
* Those who have used glucocorticoids or other immunosuppressants in the last 3 months;
* Suffering from haematological disorders such as coagulation abnormalities and thrombocytopoietic disorders;
* Those who are allergic to ultraviolet light and photosensitive treatment;
* Scar constitution;
* Those with current or previous history of skin cancer or family history of skin cancer;
* Those with infectious diseases such as HIV, syphilis, hepatitis B or C;
* Those with other serious systemic diseases;
* Patients who, in the judgement of the investigator, are not suitable for inclusion in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-10-14 (Estimated)

PRIMARY OUTCOMES:
VASI (vitiligo area severity index) score | up to 24 weeks
  The calculation of VASI (vitiligo area severity index) scores was performed by analysing standard photographs taken in the clinic at each specified follow-up time. The range is 0-100 and lower scores mean a better outcome.
VASI improvement | up to 24 weeks
  VASI improvement rate = (VASI baseline - VASI follow-up) / VASI baseline × 100 %. The range is 0-100% and higher index means a better outcome.
Side effect questionnaire and Dermatology Life Quality Index (DLQI) | up to 24 weeks
  The side effect questionnaire includes discomfort such as pain, itching, erythema, or allergic reactions. The dermatology life quality index (DLQI) range is 0-30 and higher scores mean a better outcome.

SECONDARY OUTCOMES:
Average pigmentation value, average erythema value | up to 24 weeks
  They are observed and calculated by Antera 3D.
Pigment and erythema mode images | up to 24 weeks
  They are captured by Antera 3D.
Repigmentation patterns | up to 24 weeks
  They are observed by Antera 3D.

CONTACTS AND LOCATIONS:
Overall Officials: Yijian Zhu, M.D., Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Elsaadany AE, El-Khalawany M, Elshahid AR, Seddeik Abdel-Hameed AK. Comparison between 308-nm excimer light alone versus 308-nm excimer light and platelet-rich plasma in the treatment for localized vitiligo. J Cosmet Dermatol. 2022 Jul;21(7):2826-2831. doi: 10.1111/jocd.14582. Epub 2021 Oct 31. PMID 34719101
- [Result] Deng Y, Li J, Yang G. 308-nm Excimer Laser Plus Platelet-Rich Plasma for Treatment of Stable Vitiligo: A Prospective, Randomized Case-Control Study. Clin Cosmet Investig Dermatol. 2020 Jul 23;13:461-467. doi: 10.2147/CCID.S260434. eCollection 2020. PMID 32801821
- [Result] Ibrahim ZA, El-Ashmawy AA, El-Tatawy RA, Sallam FA. The effect of platelet-rich plasma on the outcome of short-term narrowband-ultraviolet B phototherapy in the treatment of vitiligo: a pilot study. J Cosmet Dermatol. 2016 Jun;15(2):108-16. doi: 10.1111/jocd.12194. Epub 2015 Dec 23. PMID 26695436